CLINICAL TRIAL: NCT01722279
Title: The Long Term Impact of Bariatric Surgery on Quality of Life
Status: Completed | Type: Observational
Sponsor: Ascension St. Vincent Carmel Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 10070
Record Dates: First submitted 2012-11-02; First posted 2012-11-06 (Estimated); Last update posted 2012-11-06 (Estimated); Status verified 2012-11

CONDITIONS: Obesity
Keywords: bariatric surgery; long-term outcomes; obesity
MeSH Terms: conditions — Obesity | interventions — Bariatric Surgery; Gastric Bypass; Biliopancreatic Diversion; Gastroplasty

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Bariatric surgery patients, at least 5 years post-surgery: Survey participants had bariatric surgery at the St. Vincent Bariatric Center of Excellence at least 5 years before completing survey.
  Interventions: Procedure: Bariatric surgery

INTERVENTIONS:
Procedure: Bariatric surgery
  Other Names: roux-en-y gastric bypass; gastric band; biliopancreatic diversion with duodenal switch; vertical banded gastroplasty

SUMMARY:
The primary purpose of this study is to examine the breadth, nature, and factors affecting the long term changes in physical and psychological health and quality of life (QOL) following bariatric surgery. Data will be gathered via electronic survey (SurveyMonkey), postal mail, or phone, or using a standardized questionnaire expected to last 25-35 minutes. Archival data available from patient medical records will also be gathered.

DETAILED DESCRIPTION:
Information from existing databases and medical records will be used to obtain a list of phone numbers for persons who had roux-en-y bariatric surgery at the SVBCE five or more years ago at the St. Vincent Bariatric Center of Excellence (SVBCE. The interview includes scripts that the caller will use to recruit subjects in either direct conversation, in voice mail or by leaving a message. Recruitment will cease after 400 complete post pilot interviews are obtained.

The interview covers topics related to physical and psychological health and quality of life. The number of questions asked will vary from subject to subject since some questions are asked only if a prior question is answered affirmatively. For example, if a subject responds "yes" when asked "have you had plastic surgery?" the subject is then asked what type of procedure they had. The topics covered are as follows: weight, current health, post surgery complications, relationships, work, cross addiction, mental health, diet, television viewing, exercise, and life satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Bariatric surgery patients of the St. Vincent Bariatric Center of Excellence who had surgery at least 5 years before the survey was administered.

Exclusion Criteria:

* Patients having bariatric surgery at facilities other than St. Vincent Bariatric Center.
* Patients who had bariatric surgery less than 5 years before the survey period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Bariatric surgery patients of the St. Vincent Bariatric Center of Excellence who had surgery at least 5 years before the survey was administered.
Sampling Method: Non-Probability Sample
Enrollment: 414 (Actual)
Dates: Start 2010-07; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Flourishing Scale (Diener et al, 2009) | 5 or more years after bariatric surgery
Satisfaction with Life Scale (Diener et al, 1985) | 5 or more years after bariatric surgery

SECONDARY OUTCOMES:
Relationship satisfaction | At least 5 years post-surgery
Substance abuse and behavioral excesses | At least 5 years post-surgery
  Assesses presence of alcohol or other drug use problems, excessive spending, and problematic gambling
Physical Health Problems | At least 5 years post-surgery
  Assesses presence of various obesity-related health problems including diabetes, hypertension, heart disease, stroke, hich cholesterol, sleep apnea, joint pain, etc.
Weight history | At least 5 years post-surgery
  Assesses pre-surgery weight, current weight, and lowest post-surgical weight.
Satisfaction with surgery | At least 5 years post-surgery
Contact with Bariatric Center caregivers | At least 5 years post-surgery

CONTACTS AND LOCATIONS:
Overall Officials: Leslie M Schuh, PhD, Principal Investigator — St. Vincent Carmel Bariatric Center of Excellence
Locations (1):
- St. Vincent Carmel Hospital Bariatric Center of Excellence, Carmel, Indiana, United States